CLINICAL TRIAL: NCT02006966
Title: The Impact of Intraoperative Systemic Lidocaine Infusion on Chronic Postoperative Pain After Video-assisted Thoracic Surgery (VATS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2013-0693
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2016-12

CONDITIONS: Lung Cancer(Primary, Metastatic); Benign Lung Mass Requiring Operation
Keywords: Systemic lidocaine; postoperative pain; Video-assisted thoracic surgery; VATS
MeSH Terms: conditions — Neoplasm Metastasis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group L (Experimental): Intravenous lidocaine infusion group
  Interventions: Drug: Systemic intravenous lidocaine infusion
- Group C (Active Comparator): Intravenous normal saline infusion - control group
  Interventions: Drug: Normal saline infusion

INTERVENTIONS:
Drug: Systemic intravenous lidocaine infusion — In group L, intravenous lidocaine infusion(0.1mg/kg) for 10minutes after induction of anesthesia. After 10 minutes, lidocaine infusion continued at rate of 3mg/kg/hr during operation, and discontinued before move the patients to PACU.
  Arms: Group L
Drug: Normal saline infusion — In group C, the patients receive same volume of normal saline
  Arms: Group C

SUMMARY:
Systemic lidocaine infusion may improve the patients' chronic post surgical pain after video-assisted thoracic surgery

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 65 years
* ASA class 1 and 2
* Patients who are scheduled for video-assisted thoracic surgery

Exclusion Criteria:

* Allergy to local anesthetics or contraindication to use of lidocaine
* Pregnancy
* Severe cardiovascular disease
* Renal failure
* Liver failure
* Neurologic and psychologic disease
* Chronic treatment with analgesics or chronic pain patients
* Previous history of thoracic surgery (open or video-assisted)
* Patients' refusal

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08-22 (Actual); Study Completion 2016-08-22 (Actual)

PRIMARY OUTCOMES:
Assessing pain score after operation | 2 months after operation
  Assessing pain score by Short-form McGill pain questionnaire at 2 months after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea